CLINICAL TRIAL: NCT05811052
Title: The Effect of Suboccipital Release Technique on Trapezius Muscle Activation and Pain in Individuals With Anxiety
Brief Title: The Effect of Suboccipital Release Technique in Individuals With Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Sezen Tezcan, Assist. Prof, Abant Izzet Baysal University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AIBU-FTR-ST-02
Record Dates: First submitted 2023-03-20; First posted 2023-04-13 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Anxiety; Trapezius Muscle Strain; Pain
MeSH Terms: conditions — Anxiety Disorders; Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Suboccipital Release Group (Experimental)
  Interventions: Other: Suboccipital Release Technique
- Control Group (Sham Comparator)
  Interventions: Other: Sham Suboccipital Release

INTERVENTIONS:
Other: Suboccipital Release Technique — The suboccipital release technique was applied to the participants in the experimental group by an experienced practitioner who had received osteopathy training. The individual lay in the supine position, and the practitioner applied the relaxation technique by placing his hands on the patient's nape-atlantooccipital joint. The application was continued until the relaxation of the muscles under the hand of the practitioner.
  Arms: Suboccipital Release Group
Other: Sham Suboccipital Release — The participants in the control group were given a sham application by touching the hands of the therapist on the nape of the neck and waiting for a while.
  Arms: Control Group

SUMMARY:
The purpose of this study is to determine the immediate effect of the suboccipital release technique on trapezius muscle pain threshold, muscle activation, and anxiety level in individuals with anxiety.Thirty-six people with anxiety symptoms were included in the study. These people were divided into two groups, 18 control group and 18 treatment group. Upper trapezius muscle pain threshold, muscle activation and anxiety levels were evaluated. The experimental group received a single session of suboccipital release technique. The control group received a single session of sham suboccipital release. The evaluations were performed before and immediately after the treatment.The suboccipital release technique can increase the trapezius muscle upper part pain threshold and concentric muscle activation immediately after the application in individuals with anxiety.

ELIGIBILITY:
Inclusion Criteria:

* Being over the age of 18
* Agree to participate the study

Exclusion Criteria:

* Use psychiatric, analgesic and antispasmodic drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-07-06 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
The State- Trait Anxiety Inventory | Change from Baseline Anxiety Level at immediately after treatment
  The State Anxiety Scale includes questions that require the respondent to answer by taking into account his/her current feelings, while the Trait Anxiety Scale includes questions that evaluate how the respondent feels in general. It is a 4-point Likert scale. The total score obtained from both scales is minimum 20 and maximum 80. A high score indicates a high level of anxiety and a low score indicates a low level of anxiety.
Pain Assessment | Change from Baseline anxiety level at Immediately After treatment
  Pain threshold was evaluated with a manual algometer device. The midpoint of the upper trapezius muscle and the tender point with the highest pain were marked.
Surface Electromyography Measurements | Change from Baseline anxiety level at Immediately After treatment
  Maximum Voluntary Concentration (MVC) value was then measured. For the MVC value, individuals were asked to push their shoulders up (in the upward direction) against a manual resistance for 5 seconds. The measurement was repeated 3 times and 2 rests were taken after each measurement. The highest of the values was used for normalization. Afterwards, the subjects were asked to perform active shoulder elevation (concentric activity) for 3 seconds and return to neutral position for 3 seconds with the metronome. For normalization, % MVC and function % MVC values were calculated using the values recorded for all recordings.
Hospital Anxiety and Depression Scale | Baseline
  Toplam 14 maddeden oluşan (/ Anksiyete ve 7 Depresyon sorusu). 4'lü Likert tipinde bir ölçektir. 0-3 arasında bir puanlama yapılırç 0-1 puan hasta olmayan, 2 puan sınırda hasta, 2-3 puan ağır hasta olarak değerlendirilir.

SECONDARY OUTCOMES:
Cranial Rhythm | Change from Baseline anxiety level at Immediately After treatment
  Individuals were placed on the treatment bed in the supine position. The therapist touched the individual's skull and recorded the number of cycles received in one minute.

CONTACTS AND LOCATIONS:
Locations (1):
- sezen Tezcan, Bolu, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No